CLINICAL TRIAL: NCT04864574
Title: Childcare Outdoor Learning Environments as Active Food Systems: Effectiveness of the Preventing Obesity by Design (POD) Gardening Component
Brief Title: Childcare Outdoor Learning Environments as Active Food Systems
Acronym: COLEAFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Carolina State University (Other)
Responsible Party: Principal Investigator, Nilda Graciela Cosco, Principal Investigator, North Carolina State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-68001-26354 NIFA
Record Dates: First submitted 2021-04-10; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Pediatric Obesity; Sedentary Behavior
Keywords: Childhood obesity; Gardening; Fruit consumption; Vegetable consumption
MeSH Terms: conditions — Pediatric Obesity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Childcare centers were randomly assigned to one of three groups: Group 1, intervention (5 centers); Group 2, wait list control (5 centers); Group 3, no-intervention control (5 centers).
  In Year 1 (Spring), baseline data was collected from Groups 1 and 2. Group 1, initial intervention centers, received the garden intervention in the summer of Year 1 and both groups were assessed in the Fall, post intervention. No further data was collected from Group 1.
  In Year 2, Groups 2 and 3 were assessed in the Spring. Group 2, the wait-list control centers, received the garden intervention in the summer of Year 2, and both Groups 2 and 3 were assessed in the Fall of Year 2.
  No further data was collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 - Intervention (Experimental): Participating children have daily access to the fruit and vegetable garden beginning Year 1.
  Interventions: Other: Garden installation
- Group 2 - Wait-list control (delayed intervention) (Experimental): Participating children have daily access to the fruit and vegetable garden beginning Year 2.
  Interventions: Other: Garden installation
- Group 3 - Control (No Intervention): No intervention

INTERVENTIONS:
Other: Garden installation — Garden installation: 6 raised planting beds (4x6x16") configured in a single line with direct sun at least 6 hrs./day, close to hose bib, sufficient distances to allow working from most sides, vegetable vines spill over space, and storage unit for tools.
  Planting beds constructed from a standard kit. Beds filled with high quality growing medium.
  Plants selection criteria: a) documented harvest success in NC Piedmont; b) able to be eaten raw, c) harvest times at the same time (except strawberries).
  Designated beds and plants: Bed 1: 4 pepper, 2 tomato; Bed 2: 20 bean on 2 mini-teepees, 2 cucumber (trellised); Bed 3: 1 yellow squash, 1 zucchini; Bed 4: 2 blueberry bushes, 12 strawberry; Bed 5: 2 cantaloupe. Bed 6: 2 watermelon. 2 Blackberries planted at ground level on trellis.
  Arms: Group 1 - Intervention; Group 2 - Wait-list control (delayed intervention)

SUMMARY:
The aim of this project is to assess the effectiveness of the fruit and vegetable (FV) gardening component of the Preventing Obesity by Design strategy to support preschool fresh fruit and vegetable knowledge, liking and consumption, and physical activity in children 3-5 years old living in under-resourced communities and attending childcare using a Randomized Controlled Trial research design. Sample: 15 childcare centers, 286 children.

DETAILED DESCRIPTION:
Objective: To assess the effectiveness of a gardening component on preschool children's knowledge, liking and consumption of fruit and vegetable consumption, and their level of physical activity during gardening season.

Intervention: Fruit and vegetable garden installation. Childcare centers were randomly assigned to one of three groups: Group 1, intervention (5 centers); Group 2, wait list control (5 centers); Group 3, no-intervention control (5 centers).

In Year 1 (Spring), baseline data was collected from Groups 1 and Group 2 (waitlist). Group 1, initial intervention centers, received the garden intervention in the Summer and both groups were assessed in the Fall, post intervention. No further data was collected from Group 1.

In Year 2 (Spring), Group 2 (waitlist, now intervention) and Group 3 were assessed. Group 2, received the garden intervention in the Summer of Year 2 and both groups were assessed in the Fall of Year 2.

No further data was collected.

Sample: 15 centers. Children: 286 (4 and 5 years old). Center demographic profile includes child data: age, gender, parental education, race/ethnicity, special needs, and height/weight (BMI). To avoid losing "graduating" five year old children, post-intervention data was gathered before school start date.

ELIGIBILITY:
Inclusion Criteria:

* Children enrolled in selected childcare centers
* Parental consent
* Child consent to participate at the time of data collection

Exclusion Criteria:

* No parental consent

Ages: 42 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 286 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Change in mean fruit knowledge 6-item, measured by pictorial questionnaire after 5 months of gardening. | Change from baseline to 5 months
  Measured by presenting child with an image of each of 6 fruit on a tablet screen and asking the child if he/she knows (Y/N) the fruit. Pictorial questionnaire based on Carraway-Stage, V., Spangler, H., Borges, M., & Goodell, L. S. (2014). Evaluation of a pictorial method to assess liking of familiar fruits and vegetables among preschool children. Appetite, 75, 11-20.
  Six fruits: apple, blueberries, blackberry, strawberry, cantaloupe, watermelon. Same fruits were planted in the garden except for apple that takes too long to produce fruit
Change in mean vegetable knowledge 6-item, measured by pictorial questionnaire after 5 months of gardening. | Change from baseline to 5 months
  Measured by presenting child with an image of each of 6 vegetables on a tablet screen and asking the child if he/she knows (Y/N) the vegetable. Pictorial questionnaire based on Carraway-Stage, V., Spangler, H., Borges, M., & Goodell, L. S. (2014). Evaluation of a pictorial method to assess liking of familiar fruits and vegetables among preschool children. Appetite, 75, 11-20.
  Six vegetables: cucumber, green bean, red pepper, yellow squash, tomato, and zucchini. Same vegetables were planted in the garden.
Change in mean fruit liking 6-item, measured by 5-point scale pictorial questionnaire after 5 months of gardening. | Change from baseline to 5 months
  Measured by presenting child with an image of each of the 6 fruit (one by one) on a tablet screen and asking she/he to indicate whether the fruit is super yummy, yummy, just okay, yucky, super yucky by pointing at one of 5 non-gendered faces representing a 5-point scale of liking. This age-appropriate measure is based upon Carraway-Stage, V., Spangler, H., Borges, M., & Goodell, L. S. (2014). Evaluation of a pictorial method to assess liking of familiar fruits and vegetables among preschool children. Appetite, 75, 11-20.
  Six fruits: apple, blueberries, blackberry, strawberry, cantaloupe, watermelon. Same fruits were planted in the garden except for apple that takes too long to produce fruit.
Change in mean vegetable liking 6-item, measured by 5-point face scale pictorial questionnaire after 5 months of gardening. | Change from baseline to 5 months
  Measured by presenting child with an image of each of the 6 vegetables (one by one) on a tablet screen and asking she/he to indicate whether the vegetable is super yummy, yummy, just okay, yucky, super yucky by pointing at a one of 5 non-gendered faces representing a 5-point scale of liking. This age-appropriate measure is based upon Carraway-Stage, V., Spangler, H., Borges, M., & Goodell, L. S. (2014). Evaluation of a pictorial method to assess liking of familiar fruits and vegetables among preschool children. Appetite, 75, 11-20.
  Six vegetables: cucumber, green bean, red pepper, yellow squash, tomato, and zucchini. Same vegetables were planted in the garden.
Change in fruit consumption, measured by mean weight of 6 snack-time fruit consumed after 5 months of gardening | Change from baseline to 5 months
  Objective measurement of grams of fruit consumed during snack time data collection. Store-bought, standard pieces of fruits offered on individual segmented trays (6" x 12"). Each tray is labeled with a child's ID number. Six fruits (approximately 50gr/each are served). The measure is based on the Fruit & Vegetable Snack Tool, Witt KE, Dunn C. Increasing Fruit and Vegetable Consumption among Preschoolers: Evaluation of Color Me Healthy. J Nutr Educ Behav. 2012;44(2):107-113.
  Fruit servings are weighed in grams before and after the snack consumption session to the nearest .01gr. Fruits offered for consumption are the same as shown on pictorial tablet questionnaires (knowledge and liking) and planted in the intervention gardens except for apple that takes too long to produce fruit.
  Six fruits: apple, blueberries, blackberry, strawberry, cantaloupe, watermelon.
Change in vegetable consumption, measured by mean weight of six snack-time vegetables consumed after 5 months of gardening | Change from baseline to 5 months
  Objective measurement of grams of vegetable consumed during snack time data collection. Store-bought, standard pieces of vegetables offered on individual segmented trays (6" x 12"). Each tray is labeled with a child's ID number. Six vegetables (approximately 50gr/each) are served. The measure is based on the Fruit & Vegetable Snack Tool, Witt KE, Dunn C. Increasing Fruit and Vegetable Consumption among Preschoolers: Evaluation of Color Me Healthy. J Nutr Educ Behav. 2012;44(2):107-113.
  Vegetable servings are weighed in grams before and after the snack consumption session to the nearest .01gr. Vegetables offered for consumption are the same shown on pictorial tablet questionnaires (knowledge and liking) and planted in the intervention gardens.
  Six vegetables: cucumber, green bean, red pepper, yellow squash, tomato, and zucchini.
Change in physical activity level (percent of day at sedentary, moderate, and vigorous levels), measured by Actigraph GT3x+ after 5 months of gardening activities. | Change from baseline to 5 months
  Children wear Actigraph GT3x+ accelerometers for three consecutive days during same weeks of Outcome 1 - 6 data collection in April (before garden installation) and August (end of garden season) each study year.
  Minutes of sedentary (< 8.3 counts/5 sec), light (8.4-191 counts/5 sec), moderate (192-334 counts/5 sec), and vigorous (≥335 counts/5 sec) physical activity is computed based on METS.
  The measure is based on Evenson KR, Catellier DJ, Gill K, Ondrak KS, McMurray RG. Calibration of two objective measures of physical activity for children. J Sports Sci. 2008;26(14):1557-1565. doi:10.1080/02640410802334196

CONTACTS AND LOCATIONS:
Overall Officials: Nilda G Cosco, PhD, Principal Investigator — NC State University, College of Design
Locations (15):
- United States (15):
  - White Plains Children's Center, Cary, North Carolina
  - The Goddard School, Cary, North Carolina
  - Kiddie Academy of Fuquay, Fuquay-Varina, North Carolina
  - Ready or Not, Here I Grow, Fuquay-Varina, North Carolina
  - Kids Educational Center, Knightdale, North Carolina
  - Touched by an Angel Open Arms, Knightdale, North Carolina
  - La Petite Academy - Leesville, Raleigh, North Carolina
  - KinderCare Learning Center, Raleigh, North Carolina
  - La Petite Academy - Hedingham, Raleigh, North Carolina
  - Raleigh Rainbow Child Care Center, Raleigh, North Carolina
  - Appletree Child Development Center, Inc. #3, Raleigh, North Carolina
  - Kids First Academy, Raleigh, North Carolina
  - Kreepers N Krawlers Child Care Center, Raleigh, North Carolina
  - Appletree Child Development Center, Inc. #4, Raleigh, North Carolina
  - The Learning Experience, Wake Forest, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
The Study Protocol and Statistical Analysis Plan (SAP) will shared at the the end of the study after results and conclusion have been published.
Supporting Information: Study Protocol, SAP
Time Frame: Six months after publication
Access Criteria: Selected data will be shared via corresponding authors of scientific articles.
  Corresponding authors will review requests and release Study Protocols and Statistical Plan as appropriate.

REFERENCES:
- [Derived] Cosco NG, Wells NM, Zhang D, Goodell LS, Monsur M, Xu T, Moore RC. Hands-on childcare garden intervention: A randomized controlled trial to assess effects on fruit and vegetable identification, liking, and consumption among children aged 3-5 years in North Carolina. Front Psychol. 2022 Nov 10;13:993637. doi: 10.3389/fpsyg.2022.993637. eCollection 2022. PMID 36438334